CLINICAL TRIAL: NCT04436341
Title: Epileptic Activity in Patients With Alzheimer's Disease and Lewy Body Dementia
Acronym: AD-LBD-EPI
Status: Completed | Type: Observational
Sponsor: Danish Dementia Research Centre (Network)
Collaborators: Zealand University Hospital (Other); Rigshospitalet, Denmark (Other); University of Aarhus (Other); T&W Engineering A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: H-17035751
Record Dates: First submitted 2019-09-28; First posted 2020-06-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Lewy Body Disease; Epilepsy
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — A total of 13 mL of blood will be collected from each participant. Afterwards, the blood will be centrifuged and the serum, plasma and the white blood cells will be extracted. These samples will be stored in the Danish Dementia Biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Alzheimer's disease: No treatment interventions. Investigations: physical examination, ear EEG, cranial MR, cognitive tests, blood samples
- Patients with Lewy body dementia: No treatment interventions. Investigations: physical examination, ear EEG, cranial MR, cognitive tests, blood samples
- Healthy controls: No treatment interventions. Investigations: physical examination, ear-EEG cranial MR, cognitive tests, blood samples

SUMMARY:
In the current study, the investigators will examine the extent of subclinical epileptic activity in patients with Alzheimer's disease and patients with Lewy body dementia as compared to healthy elderly controls. The participants will wear a new device called "ear-EEG", which makes it possible to record EEG for longer periods of time while at home. Furthermore, the investigators want to investigate whether there is an association between subclinical epileptic activity and the cerebral blood flow as measured with functional MRI.

ELIGIBILITY:
Inclusion Criteria (Alzheimer's disease):

* Meet the criteria for probable Alzheimer's disease with amnestic presentation as described in the NIA-AA criteria (McKhann 2011)
* The diagnosis has been made by either a neurologist, psychiatrist or a geriatrician at the memory clinic at Rigshospitalet or Zealand University Hospital
* The participant is between 50 and 90 years old
* The MMSE score is between 16-28
* The participant does not wear a hearing aid
* The participant is a native Danish speaker
* The participant has at least attended school for 7 years
* The participants' hearing and vision is sufficient to participate in neuropsychological tests
* The participants' general condition of health allows that the participant can cooperate with the trial
* The participant does not suffer from psychiatric diseases (except mild depressive symptoms or mild depression) or neurological diseases that affect the brain other than Alzheimer's disease
* The treatment with anti-dementia medication or SSRI drugs have been given in stable dose for at least 3 months up to the inclusion and the doctor including the participant estimates that treatment will not change within the next 6 months
* No overuse of alcohol or intake of illegal drugs within the last 2 years
* The participant has previously undergone a CT or MRI scan, which is compatible with Alzheimer's disease
* The participant does not have any contraindications for MRI or MRI contrast
* The participant is living with another person, who is willing to take part in the trial, and who is together with the person long enough to observe the behavior (if any epileptic activity should arise)

Exclusion Criteria (Alzheimer's disease):

* Diagnosis of epilepsy prior to the diagnosis of Alzheimer's disease was made
* Other focal pathology in the hippocampus for example hippocampal sclerosis
* The person living with the participant is not able to participate (e.g. due to a serious disease or disability) in the clinical visits or able to register behavior suspected of epilepsy
* The participant is living in a nursing home
* The participant is treated with antiepileptic medication, tricyclic antidepressants or antipsychotics
* Daily or nearly daily intake of medication known to have an anticholinergic or an adrenergic effect, which is suspected to affect the cognitive abilities or the EEG
* Large brain infarctions or more than 4 lacunar infarcts
* The participants is suffering from uncontrollable movements of the face as for example oral dyskinesia

Inclusion Criteria (Lewy body dementia):

* Meet the criteria for Lewy body dementia as described in dementia with Lewy body consortium (McKeith 2017)
* The diagnose has been made by either a neurologist, psychiatrist or a geriatrician at the memory clinic at Rigshospitalet or Zealand University Hospital
* The participant is between 50 and 90 years old
* The MMSE score is between 16-28
* The participant does not wear a hearing aid
* The participant is a native Danish speaker
* The participant has at least attended school for 7 years
* The participants' hearing and vision is sufficient to participate in neuropsychological tests
* The participants' general condition of health allows that the participant can cooperate with the trial
* The participant does not suffer from psychiatric diseases (except mild depressive symptoms or mild depression) or neurological diseases that affect the brain other than Lewy body dementia
* The treatment with anti-dementia medication or SSRI drugs have been given in stable dose for at least 3 months up to the inclusion and the doctor including the participant estimates that treatment will not change within the next 6 months
* No overuse of alcohol or intake of illegal drugs within the last 2 years
* The participant does not have any contraindications for MRI or MRI contrast
* The participant is living with another person, who is willing to take part in the trial, and who is together with the person long enough to observe the behavior (if any epileptic activity should arise)

Exclusion Criteria (Lewy body dementia):

* Diagnosis of epilepsy prior to the diagnosis of Lewy body dementia was made
* Other focal pathology in the hippocampus for example hippocampal sclerosis
* The person living with the participant is not able to participate (e.g. due to a serious disease or disability) in the clinical visits or able to register behavior suspected of epilepsy
* The participant is living in a nursing home
* The participant is treated with antiepileptic medication, tricyclic antidepressants or antipsychotics
* Daily or nearly daily intake of medication known to have an anticholinergic or an adrenergic effect, which is suspected to affect the cognitive abilities or the EEG
* Large brain infarctions or more than 4 lacunar infarcts
* The participants is suffering from uncontrollable movements of the face as for example oral dyskinesia

Inclusion Criteria (Healthy controls):

* Normal cognition as evaluated at the clinical examination
* The participant is a native Danish speaker
* The participant has at least attended school for 7 years
* The participants' hearing and vision is sufficient to participate in neuropsychological tests
* The participants' general condition of health allows that the participant can cooperate with the trial
* The participant does not suffer from psychiatric diseases (except mild depressive symptoms or mild depression) or neurological diseases that affect the brain
* The participant does not have any contraindications for MRI or MRI contrast

Exclusion Criteria (Healthy controls):

* The participants is suffering from uncontrollable movements of the face as for example oral dyskinesia
* The participant is suffering from epilepsy or receives anti-epileptic medication

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the first part of the study (feasibility), the investigators will include 10 patients with Alzheimer's disease from the memory clinics at Rigshospitalet and Zealand University Hospital - Roskilde. In the main study, the investigators will include an additional 40 patients with Alzheimer's disease, 20 patients with Lewy body dementia, and 50 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility study: Investigate whether patients with Alzheimer's disease are able wear ear-EEG for longer than 24 hours during a 48 hours period | 8 months
  If it is possible for patients with Alzheimer's disease to wear ear-EEG for at least 24 hours including 5 hours of sleep during a 48 hours period
Epileptic activity in patients with Alzheimer's disease and Lewy body dementia as compared to healthy elderly controls | 2 years
  Compare the prevalence and type of paroxysmal activity as measured with the ear-EEG in patients with Alzheimer's disease and Lewy body dementia as compared to healthy elderly controls

OTHER OUTCOMES:
The correlation between cerebral blood flow and paroxysmal acitivity | 2 years
  Compare the amount of paroxysmal activity as measured with ear-EEG and the cerebral blood flow (rCBF) as measured with arterial spin labeling fMRI in patients with Alzheimer's disease and Lewy body dementia

CONTACTS AND LOCATIONS:
Overall Officials: Gunhild Waldemar, MD, Principal Investigator — Danish Dementia Research Centre; Christian S Musaeus, MD, Principal Investigator — Danish Dementia Research Centre; Troels W Kjær, MD, Principal Investigator — Zealand University Hospital - Roskilde; Kristian S Frederiksen, MD, Principal Investigator — Danish Dementia Research Centre
Locations (2):
- Denmark (2):
  - Gunhild Waldemar, Copenhagen, Copenhagen OE
  - Troels Wesenberg Kjær, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Musaeus CS, Kjaer TW, Lindberg U, Vestergaard MB, Bo H, Larsson W, Press DZ, Andersen BB, Hogh P, Kidmose P, Hemmsen MC, Rank ML, Hasselbalch SG, Waldemar G, Frederiksen KS. Subclinical epileptiform discharges in Alzheimer's disease are associated with increased hippocampal blood flow. Alzheimers Res Ther. 2024 Apr 12;16(1):80. doi: 10.1186/s13195-024-01432-9. PMID 38610005

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT04436341/Prot_SAP_000.pdf